CLINICAL TRIAL: NCT00940602
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trial of Deferasirox in Patients With Myelodysplastic Syndromes (Low/Int-1 Risk) and Transfusional Iron Overload
Brief Title: Myelodysplastic Syndromes (MDS) Event Free Survival With Iron Chelation Therapy Study
Acronym: TELESTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CICL670A2302; 2009-012418-38 (EudraCT Number)
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: TELESTO; MDS Study; Myelodysplastic Syndromes; Myelodysplastic Syndromes (low-int-1 risk)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Deferasirox

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients, investigator staff, persons performing the assessments, and data analysts remained blind to the identity of the study treatment from the time of randomization until database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deferasirox (Experimental): 10 mg/kg/day (once daily) for the first 2 weeks of treatment, followed by 20 mg/kg/day (once daily) from Week 2 to End of Treatment. After 3 months of treatment at 20 mg/kg/day, the dose was allowed to be adjusted by 5 or 10 mg/kg/day up to 40 mg/kg/day based on serum ferritin responses. When a target serum ferritin level was reached (usually between 500 and 1000 µg/L), the dose could be reduced by 50% to maintain the serum ferritin within the target range.
  Interventions: Drug: Deferasirox
- Placebo (Placebo Comparator): 10 mg/kg/day (once daily) for the first 2 weeks of treatment, followed by 20 mg/kg/day (once daily) from Week 2 to End of Treatment. After 3 months of treatment at 20 mg/kg/day, the dose was allowed to be adjusted by 5 or 10 mg/kg/day up to 40 mg/kg/day based on serum ferritin responses. When a target serum ferritin level was reached (usually between 500 and 1000 µg/L), the dose could be reduced by 50% to maintain the serum ferritin within the target range.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deferasirox — Deferasirox provided as 125 mg, 250 mg, and 500 mg dispersible tablets for oral use
  Other Names: ICL670, Exjade®
  Arms: Deferasirox
Drug: Placebo — Inactive ingredients used as a placebo comparator, provided as 125 mg, 250 mg, and 500 mg dispersible tablets for oral use
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind trial to evaluate deferasirox vs placebo in patients with myelodysplastic syndromes (low/int-1 risk) and transfusional iron overload .The trial was conducted in 17 countries, started in 2010 and ended in 2018.

DETAILED DESCRIPTION:
This randomized, double blind trial to evaluate deferasirox vs placebo in patients with myelodysplastic syndromes (low/int-1 risk) and transfusional iron overload consisted of four periods, a screening period, a treatment period, a post treatment follow-up period and a survival period. The trial recruitment period lasted until December 2014 and the trial continued for three years from the date the last patient enrolled until February 2018 (last patient last visit date).

Screening period:

The screening period lasting up to 35 days with two screening visits, at least 14 days apart, used to assess patient eligibility. Eligible patients with low or int-1 risk myelodysplastic syndromes (MDS) with transfusional iron overload were randomized in a 2:1 ratio to deferasirox or placebo respectively. Randomization was also stratified using the International prognostic scoring system of low or int-1 MDS and by geographical region (Asian vs non-Asian countries) since the Asian population has been reported to have a longer survival.

The following concomitant medications could be permitted for use while the patient was on study, and information outlining start date(s) and end date(s) of each medication taken were to be recorded on the appropriate eCRF: Erythropoietin (growth factor), G-CSF (growth factor), GM-CSF growth factor), Azacitidine, Thalidomide, Arsenic trioxide, Lenalidomide, Decitabine, Cyclosporine A, Vitamin C supplements (≤ 200 mg/day)

Treatment period:

The dosing schedule was 10 mg/kg/day (once daily) for the first 2 weeks, followed by 20 mg/kg/day (once daily). After 3 months of treatment at the dose of 20mg/kg/day, the dose could be adjusted by 5 or 10 mg/kg/day up to 40 mg/kg/day based on the serum ferritin response. Placebo matching to each strength of the active deferasirox was utilized to maintain the double-blind trial design.

During the treatment period patients returned to the investigational site every four weeks for routine procedures and to monitor safety, efficacy and compliance to treatment.

An external Data Monitoring Committee (DMC) monitored patient safety and trial conduct and received a blinded summary of serious adverse events.

All suspected endpoint events were reviewed and adjudicated by the Endpoint Adjudication Committee (EAC) to ensure that all events that were reported were judged uniformly using the same criteria. The first confirmed suspected endpoint event for a patient was counted for the trial's composite primary endpoint, "event free survival". The composite primary endpoint, "event free survival," was defined for a patient as the date randomized to trial treatment to the date of the first documented non-fatal event, related to cardiac and liver function, transformation to AML, or death due to any cause.

When a patient had a non-fatal event, related to cardiac and liver function, and transformation to AML, the trial treatment (deferasirox or placebo) was discontinued. After trial treatment was discontinued, a 28 days post treatment safety assessment for AEs and SAEs was completed. Any patient who died during the treatment or 28 day post treatment safety assessment is represented in the all-cause mortality table in the safety section of this result. After trial treatment was discontinued for a patient, their treatment was un-blinded. Subsequent iron chelation treatment was subject to the patient's and investigator's decision. Patients continued to be followed during the post-treatment evaluation or survival follow up period, depending on their choice.

For patients who did not meet a non-fatal event, study treatment was continued as long as the patient and the treating physician felt it was in the best interest for the patient or until the trial terminated/completed. There was no un-blinding of the trial treatment for patients who terminated trial treatment without meeting a non-fatal event. Patients continued to be followed during the post-treatment evaluation or survival follow up period, depending on their choice.

A patient who discontinued study treatment without meeting a non-fatal component of the composite primary endpoint continued to be evaluated every 3 months. Once a patient stopped study evaluations they were followed for at least every 6 months for overall survival and any iron chelation therapies they are receiving up to the end of study.

Post-treatment evaluation period:

For patients who had a non-fatal event: After treatment termination, all patients were followed for safety (28 days) and then evaluated with visits every three months if they agreed to move into the post treatment evaluation phase.

For patients who did not meet a non-fatal event: After termination of study treatment, if a patient and investigator chose the post-treatment evaluation period, the patient was followed for safety and endpoints at visits occurring every three months.

Survival Follow Up period:

Subsequent to the post treatment evaluation period, or at the end of treatment period, if a patient and treating physician decided that the patient would not participate in the post treatment evaluation period, the patient was followed every 6 months for overall survival and iron chelation therapies.

The end of the study was defined as three years from the date the last patient was enrolled (last patient first visit).

The sample size of 210 patients did not provide sufficient power for testing statistical hypotheses. The statistical analysis was revised accordingly to concentrate on evaluating the treatment effect of deferasirox relative to placebo, and the study phase designation was changed from Phase lll to Phase II. Amendment 4 of the study adjusted the sample size, statistical analysis, and duration of the study and added two secondary endpoints: Hematologic improvement (HI) in terms of erythroid response and Frequency and rate of infections requiring intravenous (IV) antimicrobials. Upon approval of the amendment, patients signed a new consent form and continued the appropriate visit schedule.

ELIGIBILITY:
Inclusion Criteria:

* Weigh between 35-135 kilograms
* Low or int-1 risk MDS
* Ferritin >1000 micrograms/liter at screening
* History of transfusion of 15 to 75 Packed Red Blood Cells (PRBC) units
* Anticipated to be transfused with at least 8 units of PRBCs annually during the study
* Women of child-bearing potential using effective methods of contraception during dosing of study treatment

Exclusion Criteria:

* More than 6 months of cumulative ICT (such as daily deferasirox (Exjade®) or deferiprone or 5×/week deferoxamine)
* More than 3 years since patient began receiving regular transfusions (2 units per 8 weeks or 4 units received in a 3 month period)
* Significant proteinuria
* History of hospitalization for congestive heart failure; other heart conditions as specified in the protocol
* Systemic diseases which would prevent study treatment
* Hepatitis B; Hepatitis C; HIV
* Liver cirrhosis
* Pregnant, or breast-feeding patients, or patients of child-bearing potential not employing an effective method of birth control
* History of drug or alcohol abuse within the 12 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-03-22 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (67):
- United States (11):
  - Pacific Cancer Medical Center, Inc. PAC Center, Anaheim, California
  - Rocky Mountain Cancer Centers RMCC, Greenwood Village, Colorado
  - Willis-Knighton Cancer Center Dept of Onc, Shreveport, Louisiana
  - Henry Ford Hospital Henry Ford, Detroit, Michigan
  - Midwest Cancer Care Physicians MMCC, Kansas City, Missouri
  - Mercy Medical Research Institute SC, Manchester, Missouri
  - Glacier View Research Institute - Cancer SC, Kalispell, Montana
  - Hackensack University Medical Center Department of Research, Hackensack, New Jersey
  - University of Texas MD Anderson Cancer Center Dept of MD Anderson (16), Houston, Texas
  - Cancer Care Centers of South Texas HOAST CCC of So.TX- MedicalCenter(2), San Antonio, Texas
  - Swedish Cancer Institute Ballard Campus, Seattle, Washington
- Novartis Investigative Site, Herston, Queensland, Australia
- Bulgaria (3):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (5):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, St. Catharines, Ontario
  - Novartis Investigative Site, Québec, Quebec
- China (10):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Hong Kong (2):
  - Novartis Investigative Site, Shatin, New Territories, Hong Kong
  - Novartis Investigative Site, Hong Kong
- Italy (8):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Orbassano, TO
- Malaysia (2):
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Selangor
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- New Zealand (2):
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov-on-Don
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Zurich
- Thailand (3):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- United Kingdom (9):
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Macclesfield
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Angelucci E, Li J, Greenberg P, Wu D, Hou M, Montano Figueroa EH, Rodriguez MG, Dong X, Ghosh J, Izquierdo M, Garcia-Manero G; TELESTO Study Investigators. Iron Chelation in Transfusion-Dependent Patients With Low- to Intermediate-1-Risk Myelodysplastic Syndromes: A Randomized Trial. Ann Intern Med. 2020 Apr 21;172(8):513-522. doi: 10.7326/M19-0916. Epub 2020 Mar 24. PMID 32203980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 patient rand. to deferasirox arm did not receive study drug & was excl. from the Safety set. Terminated by Sponsor: Patients who had completed at least 3 years of on-treatment period including 28-day follow-up & were still on trial when end-of-study definition (3 years after LPFV) was reached & therefore, the study was terminated as per protocol
Pre-assignment Details: The planned sample size of 210 patients randomized in a ratio of 2:1 in favor of deferasirox was based on the feasibility of enrolling the patients and consultations with the Health Authorities.
Period: Overall Study
Arm/Group | Deferasirox | Placebo
Started (All patients to whom study treatment had been assigned by randomization (Full Analysis Set).) | 149 | 76
Safety Analysis Set (All randomized patients who received at least one dose of study medication) | 148 | 76
Full Analysis Set (All patients to whom study treatment had been assigned by randomization) | 149 | 76
Treated (Treated = Received study drug) | 148 | 76
Untreated (Untreated = Did not receive study drug) | 1 | 0
Completed | 0 | 0
Not Completed | 149 | 76
Not completed — Administrative problems | 1 | 1
Not completed — Patient/guardian decision | 13 | 28
Not completed — Physician Decision | 8 | 5
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Deviation (untreated) | 1 | 0
Not completed — Disease progression | 8 | 2
Not completed — Death | 38 | 19
Not completed — Lost to Follow-up | 3 | 1
Not completed — Patient withdrew consent | 26 | 13
Not completed — Adverse Event | 7 | 2
Not completed — Study terminated by Sponsor = trial was to continue for 3 years from date the last patient enrolled | 43 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferasirox | Placebo | Total
Number analyzed (Participants) | 149 | 76 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (16.13) | 60.7 (15.05) | 61.0 (15.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 32 | 88
  Male | 93 | 44 | 137
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/latino | 14 | 5 | 19
  Chinese | 61 | 29 | 90
  Mixed ethnicity | 1 | 0 | 1
  Other | 73 | 42 | 115
MDS risk category [Number; unit: participants] — International Prognostic Scoring System (IPSS}
  participants
    Low (combined score 0) | 41 | 21 | 62
    Intermediate 1 (combined score 0.5 - 1.0) | 108 | 55 | 163

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Event-free survival was defined as the time from the date of randomization to the date of the first documented non-fatal event (worsening cardiac function, hospitalization for congestive heart failure, liver function impairment, liver cirrhosis, transformation to AML, as defined in the protocol), or death, whichever occurred first. Participants who did not experience a non-fatal event as of the time of data cut-off (end of study), as well as participants who did not experience a non-fatal event and stopped study participation before the data cut-off, were censored as specified in the protocol.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: FAS: the FAS comprised all patients to whom study treatment had been assigned by randomization. According to the intention to treat principle, patients were analyzed according to the study treatment and strata they were assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
days | 1440 [1167 to 1559] | 1091 [820 to 1348]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — The study was not designed for confirmatory analyses. Statistical tests were performed in an exploratory sense only; p = 0.015, Regression, Cox — Exploratory p-value is one tailed and is based on the stratified log-rank test; Hazard Ratio (HR) = 0.636, 95% CI 2-sided [0.42 to 0.96] — 95% CI was based on a Wald test from Cox model

2. Secondary Outcome: Percentage of Participants With Hematologic Improvement (HI) in Terms of Erythroid Response
Description: HI in terms of erythroid responses was assessed based on International Working Group (IWG) criteria, with improvement defined as follows:
  * Hemoglobin increase of ≥ 1.5 g/dL OR
  * Reduction of ≥ 4 RBC transfusions/8 weeks in comparison to pre-treatment values and lasting at least 8 weeks. The last hemoglobin value measured prior to randomization was used as the pre-treatment value. The last available lab assessment date was used as the cut-off date for the analysis.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
percentage of participants | 39.6 [31.4 to 47.6] | 27.6 [16.9 to 38.3]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — 100 (1-α)% confidence intervals with α of 0.05 are provided; Wilson score test = 12.0, 95% CI 2-sided [-1.8 to 25.7]

3. Secondary Outcome: Overall Survival
Description: Overall survival was calculated as the date of death (irrespective of cause) minus date of randomization plus 1.
Time Frame: Day 1 to end of treatment period, approx. 7.4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
days | 1907 [1440 to NA] — NA = Not evaluable as insufficient number of events | 1509 [1095 to 1804]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — The study was not designed for confirmatory analyses. Statistical tests were performed in an exploratory sense only; p = 0.200, Regression, Cox; Hazard Ratio (HR) = 0.832, 95% CI 2-sided [0.54 to 1.28] — 95% CI was based on a Wald test from Cox model

4. Secondary Outcome: Percentage of Participants With Newly Occurring Hypothyroidism Compared to Baseline
Description: As assessed by annual measurement of Thyroid Stimulating Hormone (TSH) and free T4. Hypothyroidism was defined as follows and is inclusive of:
  * Primary hypothyroidism: serum TSH >upper limit of normal (ULN) and free T4 <lower limit of normal (LLN);
  * Secondary hypothyroidism: serum TSH <ULN and free T4 <lower limit of normal;
  * Subclinical hypothyroidism: TSH >ULN and a free T4 within normal limits. The last available lab assessment date was used as the cut-off date for the analysis.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
percentage of participants | 5.4 [1.4 to 9.3] | 3.9 [0.0 to 9.0]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — 100 (1-α)% confidence intervals with α of 0.05 are provided; Wilson score test = 1.4, 95% CI 2-sided [-5.3 to 8.1]

5. Secondary Outcome: Percentage of Participants With Worsening Glucose Metabolism Compared to Baseline
Description: As assessed by an annual glucose tolerance test (OGTT). Worsening glucose metabolism was defined as an increase in glucose metabolism category (normal, impaired glucose metabolism, diabetes mellitus) based on the American Diabetes Association criteria (American Diabetes Association 2009) compared to the baseline result. The last available lab assessment date was used as the cut-off date for the analysis.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
percentage of participants | 18.1 [11.6 to 24.6] | 18.4 [9.0 to 27.8]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — 100 (1-α)% confidence intervals with α of 0.05 are provided; Wilson score test = -0.3, 95% CI 2-sided [-12.0 to 11.4]

6. Secondary Outcome: Time to Disease Progression
Description: Disease progression was defined as follows:
  * MDS progression: Transition into a higher MDS risk group based on IPSS scoring
  * Progression to AML: 20 percent or more blasts seen in the bone marrow collected by biopsy or aspirate.
  Disease progression was calculated as follows: Date of diagnosis of MDS progression or date of first diagnosis of AML, minus date of randomization plus 1. Participants who neither experienced MDS progression nor progression to AML were censored at the last contact date.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
days | NA [NA to NA] — NA = Not evaluable as insufficient number of events | NA [NA to NA] — NA = Not evaluable as insufficient number of events
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — The study was not designed for confirmatory analyses. Statistical tests were performed in an exploratory sense only; p = 0.184, Regression, Cox; Hazard Ratio (HR) = 0.725, 95% CI 2-sided [0.36 to 1.46] — 95% CI was based on a Wald test from Cox model

7. Secondary Outcome: Time to First Occurrence of Serum Ferritin Level >2 Times the Baseline Value at Two Consecutive Assessments (at Least Two Weeks Apart)
Description: Assessed by blood draw and calculated as follows: Date of first occurrence of serum ferritin >2 times the baseline value at two consecutive assessments (at least two weeks apart), minus date of randomization plus 1. Participants who did not experience such an increase were censored at the last date when serum ferritin was available.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
days | NA [NA to NA] — NA = Not evaluable as insufficient number of events | 592 [397 to 877]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — The study was not designed for confirmatory analyses. Statistical tests were performed in an exploratory sense only; p < .001, Regression, Cox; Hazard Ratio (HR) = 0.195, 95% CI 2-sided [0.11 to 0.36] — 95% CI was based on a Wald test from Cox model

8. Secondary Outcome: Time to at Least a 10% Increase From Baseline in Left Ventricular End-diastolic Internal (LVIDD) at Two Consecutive Assessments at Least Two Weeks Apart
Description: Assessed by echocardiography and calculated as follows: Date of echocardiography assessment where a minimum of 10% increase of LVIDD first occurred, minus date of randomization plus 1. Participants who did not experience such an increase were censored at the last date when LVIDD was available.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
days | NA [871 to NA] — NA = Not evaluable as insufficient number of events | NA [732 to NA] — NA = Not evaluable as insufficient number of events
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — The study was not designed for confirmatory analyses. Statistical tests were performed in an exploratory sense only; p = 0.303, Regression, Cox; Hazard Ratio (HR) = 0.871, 95% CI 2-sided [0.52 to 1.46] — 95% CI was based on a Wald test from Cox model

9. Secondary Outcome: Time to at Least a 10% Increase From Baseline in Left Ventricular Internal Systolic Diameter (LVISD) at Two Consecutive Assessments at Least Two Weeks Apart
Description: Assessed by echocardiography and calculated as follows: Date of echocardiography assessment where a minimum of 10% increase of LVISD first occurred, minus date of randomization plus 1. Participants who did not experience such an increase were censored at the last date when LVISD was available.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
days | 1179.0 [532 to NA] — NA = Not evaluable as insufficient number of events | NA [502 to NA] — NA = Not evaluable as insufficient number of events
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — The study was not designed for confirmatory analyses. Statistical tests were performed in an exploratory sense only; p = 0.389, Regression, Cox; Hazard Ratio (HR) = 1.072, 95% CI 2-sided [0.66 to 1.75] — 95% CI was based on a Wald test from Cox model

10. Secondary Outcome: Total Number of Infections Requiring Intravenous Antimicrobials
Description: The total number of infections were counted and summarized per treatment group. For this number, one participant can contribute more than one infection event. Infections were determined from the reported AEs with system organ class "Infections and infestations" and action taken "Concomitant medication taken." Antimicrobial therapy was determined from the reported concomitant medications for participants who had an infection AE. The route of administration needed to be specified as "intravenous (i.v.)". End of treatment period was defined as the treatment period plus 28 days.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: SAS: the safety set included all randomized patients who received at least one dose of study medication. Patients were analyzed according to the study treatment they actually received and the strata they were assigned. No Statistical Analysis was performed
Measure: Number; unit: infections
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 148 | 76
infections | 253 | 111

11. Secondary Outcome: Percentage of Participants With Major Gastrointestinal Bleeding
Description: Major gastrointestinal bleeding was defined as an AE that could include one of the following MedDRA preferred terms: gastric hemorrhage, gastrointestinal hemorrhage, small intestinal hemorrhage, esophageal hemorrhage, large intestinal hemorrhage, rectal hemorrhage, melaena, duodenal ulcer hemorrhage, gastric ulcer hemorrhage, peptic ulcer hemorrhage, large intestinal ulcer hemorrhage, esophageal ulcer hemorrhage, and hematochezia. The end of treatment period was defined as the treatment period plus 28 days.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: SAS: the safety set included all randomized patients who received at least one dose of study medication. Patients were analyzed according to the study treatment they actually received and the strata they were assigned.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 148 | 76
percentage of participants | 5.4 [1.4 to 9.4] | 3.9 [0.0 to 9.0]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — 100 (1-α)% confidence intervals with α of 0.05 are provided; Wilson score test = 1.5, 95% CI 2-sided [-5.2 to 8.1]

12. Secondary Outcome: Percentage of Participants With Significant Renal Dysfunction
Description: Significant renal dysfunction was defined as a serum creatinine value ≥ 2 times upper limit of normal (ULN) at two consecutive assessments at least 7 days apart
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 148 | 76
percentage of participants | 0.7 [0.0 to 2.3] | 0 [0.0 to 0.7]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — 100 (1-α)% confidence intervals with α of 0.05 are provided; Wilson score test = 0.7, 95% CI 2-sided [-1.6 to 3.0]

13. Secondary Outcome: Percentage of Participants With Newly Occurring Moderate or Severe Neutropenia
Description: Moderate or severe neutropenia was defined as neutrophil counts less than 1.0×10E9/L.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 148 | 76
percentage of participants | 27.7 [20.2 to 35.5] | 26.3 [15.8 to 36.9]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — 100 (1-α)% confidence intervals with α of 0.05 are provided; Wilson score test = 1.4, 95% CI 2-sided [-11.9 to 14.6]

14. Secondary Outcome: Percentage of Participants With Newly Occurring Severe Thrombocytopenia
Description: Severe thrombocytopenia was defined as platelets counts less than 50×10E9/L.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 148 | 76
percentage of participants | 10.1 [4.9 to 15.3] | 19.7 [10.1 to 29.3]
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — 100 (1-α)% confidence intervals with α of 0.05 are provided; Wilson score test = -9.6, 95% CI 2-sided [-20.8 to 1.6]

15. Secondary Outcome: Time to Study Drug Discontinuation Due to an AE or Laboratory Abnormality
Description: As recorded on the Study Treatment Completion electronic Case Report Form (eCRF), date and reason given.Only participants for whom the reason for stopping study medication was entered as AE or laboratory abnormality were considered. This time to event endpoint was calculated as the date of study drug discontinuation due to an AE or laboratory abnormality minus date of randomization plus 1. Participants who did not discontinue study medication due to an AE or laboratory abnormality were censored at the date of study drug discontinuation.
Time Frame: Day 1 to end of treatment period, approx. 7 years
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 148 | 76
days | NA [1486 to NA] — NA = Not evaluable as insufficient number of events | 1022 [904 to NA] — NA = Not evaluable as insufficient number of events
Statistical Analysis 1: Comparison: Deferasirox vs Placebo; Test type: Other — The study was not designed for confirmatory analyses. Statistical tests were performed in an exploratory sense only; p = 0.232, Regression, Cox; Hazard Ratio (HR) = 0.797, 95% CI 2-sided [0.43 to 1.46] — 95% CI was based on a Wald test from Cox model

16. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from FPFT up to 28 days after study drug discontinuation, for a maximum duration of 2627 days (2599 plus 28 days) (treatment duration ranged from 1 day to 2599 days). Deaths post treatment survival follow up were collected after the on treatment period, up to approx. 7.4 years. Patients who had not experienced any of the non-fatal events from the composite primary endpoint and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: 2627 days, approx. 7.4 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 149 | 76
Participants
  Total deaths | 57 | 33
  Deaths on-treatment | 24 | 10
  Deaths post-treatment survival follow up | 33 | 23

ADVERSE EVENTS:
Time Frame: On treatment deaths were collected from FPFT up to 28 days after study drug discontinuation, for a maximum duration of 2627 days (2599 plus 28 days) (treatment duration ranged from 1 day to 2599 days).
Description: Any sign or symptom that occurs during the study treatment plus 28 days post treatment
Groups:
- All Patients: Combined patients from the Deferasirox and Placebo arms
Arm/Group | Deferasirox | Placebo | All Patients
All-Cause Mortality (participants affected / at risk) | 24/148 | 10/76 | 34/224
Serious Adverse Events (participants affected / at risk) | 80/148 | 38/76 | 118/224
Other Adverse Events (participants affected / at risk) | 135/148 | 65/76 | 200/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=148) | Placebo (N=76) | All Patients (N=224)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 11 | 3 | 14
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 1
Cytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 5
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenic lesion (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2 | 7
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0 | 2
Cardiac failure (Cardiac disorders) | 3 | 1 | 4
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 1
Aural polyp (Ear and labyrinth disorders) | 1 | 0 | 1
Hypogonadism (Endocrine disorders) | 1 | 0 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 0 | 3
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 9
Gastritis (Gastrointestinal disorders) | 1 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 2 | 6
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 1 | 2
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 5 | 0 | 5
Asthenia (General disorders) | 1 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 0 | 2
Oedema (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 2 | 2
Peripheral swelling (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 14 | 5 | 19
Cholecystitis (Hepatobiliary disorders) | 3 | 0 | 3
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 2
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 1
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 1 | 2
Anal infection (Infections and infestations) | 0 | 1 | 1
Appendiceal abscess (Infections and infestations) | 2 | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2 | 3
Clostridial infection (Infections and infestations) | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 1 | 2
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 1
Groin abscess (Infections and infestations) | 2 | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 4
Lung infection (Infections and infestations) | 9 | 4 | 13
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 1
Orchitis (Infections and infestations) | 1 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 3 | 6
Respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Scrub typhus (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 6 | 2 | 8
Septic shock (Infections and infestations) | 2 | 0 | 2
Skin graft infection (Infections and infestations) | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 2 | 2
Soft tissue infection (Infections and infestations) | 1 | 0 | 1
Tongue fungal infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 6
Urinary tract infection (Infections and infestations) | 0 | 3 | 3
Urosepsis (Infections and infestations) | 1 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood creatine increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Light chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0 | 2
Cognitive disorder (Nervous system disorders) | 1 | 0 | 1
Coma (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Hemianopia homonymous (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 2 | 3
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 4
Anuria (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 2 | 3
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=148) | Placebo (N=76) | All Patients (N=224)
Anaemia (Blood and lymphatic system disorders) | 14 | 5 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 4 | 13
Vertigo (Ear and labyrinth disorders) | 8 | 4 | 12
Abdominal discomfort (Gastrointestinal disorders) | 9 | 6 | 15
Abdominal distension (Gastrointestinal disorders) | 11 | 4 | 15
Abdominal pain (Gastrointestinal disorders) | 13 | 9 | 22
Abdominal pain upper (Gastrointestinal disorders) | 12 | 9 | 21
Constipation (Gastrointestinal disorders) | 17 | 12 | 29
Diarrhoea (Gastrointestinal disorders) | 51 | 17 | 68
Dyspepsia (Gastrointestinal disorders) | 11 | 6 | 17
Gingival bleeding (Gastrointestinal disorders) | 5 | 5 | 10
Mouth ulceration (Gastrointestinal disorders) | 13 | 1 | 14
Nausea (Gastrointestinal disorders) | 23 | 10 | 33
Vomiting (Gastrointestinal disorders) | 12 | 6 | 18
Asthenia (General disorders) | 13 | 8 | 21
Fatigue (General disorders) | 21 | 12 | 33
Non-cardiac chest pain (General disorders) | 7 | 6 | 13
Oedema peripheral (General disorders) | 22 | 9 | 31
Pyrexia (General disorders) | 42 | 13 | 55
Conjunctivitis (Infections and infestations) | 2 | 4 | 6
Influenza (Infections and infestations) | 8 | 6 | 14
Lower respiratory tract infection (Infections and infestations) | 6 | 4 | 10
Nasopharyngitis (Infections and infestations) | 10 | 4 | 14
Oral herpes (Infections and infestations) | 5 | 5 | 10
Upper respiratory tract infection (Infections and infestations) | 34 | 19 | 53
Urinary tract infection (Infections and infestations) | 14 | 8 | 22
Alanine aminotransferase increased (Investigations) | 14 | 9 | 23
Blood bilirubin increased (Investigations) | 9 | 2 | 11
Blood creatinine increased (Investigations) | 37 | 1 | 38
Creatinine renal clearance decreased (Investigations) | 16 | 3 | 19
Protein urine present (Investigations) | 8 | 1 | 9
Weight decreased (Investigations) | 12 | 6 | 18
Decreased appetite (Metabolism and nutrition disorders) | 18 | 8 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 3 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 3 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 7 | 22
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 7 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 11
Dizziness (Nervous system disorders) | 19 | 6 | 25
Headache (Nervous system disorders) | 17 | 13 | 30
Insomnia (Psychiatric disorders) | 9 | 3 | 12
Proteinuria (Renal and urinary disorders) | 12 | 1 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 11 | 41
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 14
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 14
Rash (Skin and subcutaneous tissue disorders) | 16 | 8 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT00940602/SAP_000.pdf
  • Study Protocol (2014-09-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT00940602/Prot_001.pdf